CLINICAL TRIAL: NCT05655650
Title: Identifying Biomarkers in Alzheimer's Disease
Acronym: SEEDS
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Vincent Mok, Professor, Chinese University of Hong Kong
Other Study IDs: SEEDS
Record Dates: First submitted 2022-12-09; First posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Neuro-Degenerative Disease; Alzheimer Disease
Keywords: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma, blood cells
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Normal cognition: 75 subject without any of the following: subjective memory complaint and cognitive impairment base on cognitive assessments
- Subjective Cognitive Disorder: 75 subjects without cognitive impairment based on cognitive cognitive assessments but with subject memory complaint
- Mild Cognitive Impairment: 75 subjects with both subjective memory complaints and mild cognitive impairment base on cognitive assessments
- Dementia: 75 subjects with both subjective memory complaints and moderate to severe cognitive impairment base on cognitive assessments

SUMMARY:
Alzheimer's disease is a severe neurodegenerative disorder of the brain that is characterized by progressive loss of memory and cognitive decline. With the ageing population, AD is a major public health problem affecting nearly 35 million people worldwide with numbers projected to rise to 115.4 million by 2050. AD is the only cause of death among the top ten causes that has no prevention or cure . It is believed that novel treatment of AD needs to start early or even at the prodromal stage in order to be effective. Therefore, there is an urgent need to find accurate methods of early detection before patients with AD develop clinical dementia.

This study aims to identify biomarkers for AD in local Chinese population. this study hypothesizes blood-based proteomics, retinal imaging, ASL-MRP and tau PET can improve the accuracy and staging of AD.

DETAILED DESCRIPTION:
This is a cohort study. It involves baseline and 6 yearly follow ups. At baseline, all participants will go through a list of cognitive assessments, blood taking, Brain MRI scan, Brain PET scan and retinal imaging.

At the first five yearly follow ups, cognitive assessment will be performed. For the sixth yearly follow up, automatic retinal image will be performed in addition to cognitive assessment.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* [For dementia group, clinical diagnosis of "probable Alzheimer's disease" according to recommendation from the National Institute on Aging-Alzheimer's Association workgroups (NIA-AA)

Exclusion Criteria:

* Clinical diagnosis of non-AD dementia
* contraindication for MRI or PET

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: AD subjects will be recruited from neurology cognitive disorder clinic of Prince of Wales Hospital. Age match normal control will be recruited from existing normal control studies.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
The score change in Hong Kong List Learn Test (HKLLT) | Baseline, 1 year, 2 year, 3 year ,4 year ,5 year and 6 year visit after baseline visit
  The Hong Kong List Learn Test would be administered to assess the cognitive status for all group of study subjects
The score change in Montreal Cognitive Assessment Hong Kong (HK-MoCA) | Baseline, 1 year, 2 year, 3 year ,4 year ,5 year and 6 year visit after baseline visit
  The Montreal Cognitive Assessment Hong Kong would be administered to assess the cognitive status for all group of study subjects
The score change Clinical Dementia Rating (CDR) | Baseline, 1 year, 2 year, 3 year ,4 year ,5 year and 6 year visit after baseline visit
  The Clinical Dementia Rating would be administered to assess the cognitive status for all group of study subjects
Amount of amyloid β with 11C-Pittsburgh compound B | Baseline
  Positron emission tomography imaging with 11C-Pittsburgh compound B would quantify the amount of amyloid β. Amyloid β is one of the biomarkers associate Alzheimer Disease
Amount of amyloid tau with T807 tracer | Baseline
  Positron emission tomography imaging with T807 tracer would quantify the amount of tau protein. tau protein is one of the biomarkers associate with Alzheimer Disease
Amount of glucose hypometabolism | Baseline
  Positron emission tomography imaging with 18F-FDG tracer would quantify the amount of glucose hypometabolism. glucose hypometabolism is one of the biomarkers associate with Alzheimer Disease
arterial spin labeling magnetic resonance perfusion (ASL-MRP) | Baseline
  Arterial spin labeling (ASL) perfusion is a MRI technique to quantify tissue blood flow of all group of subjects
Change of Automatic Retinal Imaging | Baseline, 6th year follow up
  There is a close anatomical correlation between both the macrovascular and the microvascular blood supply to the brain and the retina, and both vascular networks share similar vascular regulatory processes. Automatic Retinal Imaging is used to investigate microcirculations in retinal

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese University of Hong Kong, Hong Kong, Hong Hong, Hong Kong